CLINICAL TRIAL: NCT06625775
Title: A Phase 1a/1b Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of BBO-10203 in Subjects With Advanced Solid Tumors (The BREAKER-101 Study)
Brief Title: Open-Label Study of BBO-10203 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TheRas, Inc., d/b/a BBOT (BridgeBio Oncology Therapeutics) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBBO10203-101; 2024-519445-29-00 (EU CTIS Number); BREAKER-101 (Other: TheRas, Inc., d/b/a BBOT (BridgeBio Oncology Therapeutics))
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor, Adult; Metastatic Breast Cancer; Advanced Breast Cancer; HER2 Mutation-Related Tumors; HER2-positive Metastatic Breast Cancer; KRAS Mutant Metastatic Colorectal Cancer; Metastatic Lung Cancer; Metastatic Colorectal Cancer; Advanced Lung Cancer; HR-positive, HER2-negative Advanced Breast Cancer; HER2-positive Advanced Breast Cancer
Keywords: BREAKER-101; BridgeBio Oncology Therapeutics; BBOT; Phase1; Phase 1a/1b; Trastuzumab; Breast; Colorectal; Non-Small Cell Lung Cancer; CRC; NSCLC; Metastatic Cancer; Advanced Cancer; HER2-positive; HR-positive; HR-positive, HER2-negative; HER2-negative
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — Trastuzumab; Fulvestrant; ribociclib; Folfox protocol; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BBO-10203 (Experimental): Participants enrolled in this cohort will receive BBO-10203 tablets orally (different dose levels will be evaluated) once daily as monotherapy. This cohort will enroll patients with HER2-positive advanced breast cancer, HR-positive HER2-negative advanced breast cancer, advanced colorectal cancer, and advanced lung cancer.
  Interventions: Drug: BBO-10203
- BBO-10203 + Trastuzumab (Experimental): Participants enrolled in this cohort will receive BBO-10203 tablets orally in combination with trastuzumab. This cohort will enroll patients with HER2-positive advanced breast cancer.
  Interventions: Drug: BBO-10203; Drug: Trastuzumab
- BBO-10203 + Fulvestrant (Experimental): Participants enrolled in this cohort will receive BBO-10203 tablets orally in combination with fulvestrant. This cohort will enroll patients with HR-positive, HER2-negative advanced breast cancer.
  Interventions: Drug: BBO-10203; Drug: Fulvestrant; Drug: Ribociclib
- BBO10203 + Fulvestrant + Ribociclib (Experimental): Participants enrolled in this cohort will receive BBO-10203 tablets orally in combination with fulvestrant and ribociclib as determined in the dose escalation. This cohort will enroll patients with HR-positive, HER2-negative advanced breast cancer.
  Interventions: Drug: BBO-10203; Drug: Fulvestrant; Drug: Ribociclib
- BBO10203 + FOLFOX + Bevacizumab (Experimental): Participants enrolled in this cohort will receive BBO-10203 tablets orally in combination with FOLFOX and bevacizumab. This cohort will enroll patients with KRAS-mutant advanced colorectal cancer.
  Interventions: Drug: BBO-10203; Drug: FOLFOX; Drug: Bevacizumab

INTERVENTIONS:
Drug: BBO-10203 — Participants will receive assigned dose of BBO-10203 orally once daily
Drug: Trastuzumab — Participants will receive trastuzumab as infusion or subcutaneous injection every 21 days
  Arms: BBO-10203 + Trastuzumab
Drug: Fulvestrant — Patients will receive Fulvestrant as an intramuscular injection every 28 days (additional dose on C1D15)
  Arms: BBO-10203 + Fulvestrant; BBO10203 + Fulvestrant + Ribociclib
Drug: Ribociclib — Patients will receive Ribociclib orally once a day (21 days on treatment, 7 days off)
  Arms: BBO-10203 + Fulvestrant; BBO10203 + Fulvestrant + Ribociclib
Drug: FOLFOX — Patients will receive FOLFOX as infusion every 14 days
  Arms: BBO10203 + FOLFOX + Bevacizumab
Drug: Bevacizumab — Patients will receive bevacizumab as infusion every 28 days
  Arms: BBO10203 + FOLFOX + Bevacizumab

SUMMARY:
First in human study to evaluate the safety, tolerability, and pharmacokinetics (PK) of BBO-10203, a PI3Kα:RAS breaker, alone and in combination with other anti-cancer agents in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multi-center Phase 1a/1b study designed to evaluate the safety, tolerability, preliminary antitumor activity, and PK of BBO-10203 as a single agent and in combination with Trastuzumab, Fulvestrant +/- Ribociclib, or FOLFOX + Bevacizumab in patients with locally advanced unresectable or metastatic (ie, advanced) solid tumors. The study includes a dose escalation phase and an expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced and unresectable or metastatic HER2-positive advanced breast cancer (aBC), HR-positive/HER2-negative advanced breast cancer, KRAS mutant advanced colorectal cancer (aCRC), or KRAS mutant advanced non-small cell lung cancer (aNSCLC)
* Measurable disease by RECIST v1.1 (except for HR-positive HER2-negative aBC where evaluable bone-only disease is permitted)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Adequate LVEF assessed by ECHO or MUGA (BBO-10203 + Trastuzumab cohorts only)
* Stable brain metastases
* Patients with HER2-positive aBC: Must have had at least 2 prior lines of anti-HER2-directed therapy. Only 1 prior line is acceptable where there is no other regionally available standard of care (SoC)
* Monotherapy Cohort patients with HR-positive, HER2-negative aBC, KRAS mutant aCRC or aNSCLC: Must have progression on, or disease recurrence after at least one line of SOC treatment or in the opinion of the investigator, would be unlikely to tolerate or derive clinically meaningful benefit from SoC therapy
* BBO-10203 + Fulvestrant combination cohort patients with HR-positive, HER2-negative aBC: confirmed PIK3CA mutation, must have been treated with a CDK4/6i
* BBO-10203 + Fulvestrant + ribociclib combination cohort patients with HR-positive, HER2-negative aBC: confirmed PIK3CA mutation, no prior systemic therapy in the aBC setting permitted
* BBO-10203 + FOLFOX + Bevacizumab combination cohort patients with KRAS mutant aCRC: One prior line of irinotecan-containing therapy for locally advanced or metastatic CRC is allowed but not required

Exclusion Criteria:

* Patients with KRAS mutant aCRC who have KRAS G12R mutation, BRAFV600E mutation, HER2amp, or dMMR/MSI-H tumors
* Patients with KRAS mutant aNSCLC who have KRAS G12R mutation, or tumors with other targetable driver mutations (eg, EGFR, anaplastic lymphoma kinase, ROS1/BRAF/RET/MET/EGFR exon20 insertion/NTRK/HER2)
* Patients with untreated and/or non-stable brain metastases

Other inclusion/exclusion criteria are specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of BBO-10203 as a single agent | Up to approximately 5 years
Percentage of patients with treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) | Up to approximately 5 years
Recommended BBO-10203 dose in combination with trastuzumab, fulvestrant +/- ribociclib, and FOLFOX + bevacizumab | Up to approximately 5 years

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) as assessed by RECIST v1.1. | Up to approximately 5 years
Duration of response (DOR) as assessed by RECIST v1.1. | Up to approximately 5 years
Progression-free survival (PFS) as assessed by RECIST v1.1 | Up to approximately 5 years
Overall survival (OS) | Up to approximately 5 years
Area under the concentration-time curve (AUC | Predose (within 30 minutes) of C1D1 until up to approximately 5 years
Maximum plasma drug concentration (Cmax) | Predose (within 30 minutes) of C1D1 until up to approximately 5 years
Time for maximum plasma drug concentration (Tmax) | Predose (within 30 minutes) of C1D1 until up to approximately 5 years
Objective response rate (ORR) as assessed by RECIST v1.1 for patients with measurable disease | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (27):
- United States (18):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Diego Moores Cancer Center, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Moffitt Cancer Center, Tampa, Florida
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Insitute, Boston, Massachusetts
  - St. Lukes Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - SCRI at Mary Crowley, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas San Antonio (UTSA), San Antonio, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Wisconsin Institute for Medical Research, Madison, Wisconsin
- Australia (2):
  - Scientia Clinical Research, Randwick, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- France (3):
  - Institut régional du Cancer de Montpellier - Val d'Aurelle, Montpellier, Occitanie
  - lnstitut de Cancérologie de l'Ouest - Site Saint-Herblain, Saint-Herblain, Pays de la Loire Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - Hospital Beata Maria Ana, Madrid, Madrid
  - Hospital Quiron Madrid - NEXT Oncology, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes